CLINICAL TRIAL: NCT00894764
Title: A Clinical and Microbiological Study of Acute Respiratory Infections in Refugee Infants Living on the Thai-Burmese Border
Brief Title: The Study of Chest Infections in Infants Living in a Refugee Camp on the Thai-Burmese Border
Acronym: ARI
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU_09-2007; Mahidol Approval: MUTM2007/036; OXTREC Approval: 031-06
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Childhood Pneumonia; Pneumococcal Carriage
Keywords: Childhood; Pneumonia; Pneumococcal; pneumococcus; Carriage
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Routine Follow Up: Monthly nasopharyngeal swab for infant. Seen during acute illness.
- Immunology: Monthly nasopharyngeal swab for mother and infant. Serum sample taken from Infant. Seen during acute illness.

SUMMARY:
This study will follow 1000 refugee infants from birth for two years. The aim of the study is to better understand why some children develop infections caused by the bacterium Streptococcus pneumoniae whilst others merely carry this organism asymptomatically at the back of the nose (in the nasopharynx). The investigators will also define which micro-organisms cause lower respiratory tract infections (e.g., pneumonia) in this population in order to implement appropriate interventions (e.g., vaccines). Infants will be reviewed monthly and a nasopharyngeal swab will be taken. A group of 250 mother-infant pairs will be studied in greater detail, to improve our understanding of the frequency and outcomes of nasopharyngeal carriage of Streptococcus pneumoniae. Monthly nasopharyngeal swabs will be collected from mothers and infants. The investigators will measure the infant immune response to Streptococcus pneumoniae carriage or disease by taking monthly blood samples. The investigators will make an assessment of the protective effect of antibodies acquired from the mother during pregnancy by taking blood from the mother and placenta at birth. An assessment of pneumococcal carriage in mothers will also be made to determine how frequently the bacterium is transmitted between family members. All lower respiratory tract infections will be documented, and the causative micro-organisms identified.

DETAILED DESCRIPTION:
This project's central hypothesis is that acute lower respiratory infections (ALRI) are a common and significant cause of morbidity and mortality in young children living in Maela refugee camp on the Thai-Burmese border, and that this is reflective of the general situation in the developing world. Therefore, we aim to define the incidence, aetiology, and outcome of acute lower respiratory infections in this population. This will focus on Streptococcus pneumoniae and the factors associated with colonisation and invasive disease.

Additional objectives are to:

1. Characterise the interaction between bacterial and viral pathogens and disease.
2. Examine the dynamics of pneumococcal nasopharyngeal carriage, including transmission of strains between infants and their mothers.
3. Determine the effect of the non-pathogenic members of the nasopharyngeal flora on colonisation with potential pathogens.
4. Examine the role of passively transferred maternal pneumococcal antibodies in subsequent pneumococcal colonisation and disease in the infant.
5. Document the development of pneumococcal antibodies in the infants over time and correlate these with pneumococcal carriage and infection episodes.
6. Determine the risk factors associated with respiratory infection.
7. Characterise the bacteria causing invasive non-respiratory infections.
8. Conduct surveillance for influenza and in particular avian influenza A (H5N1) infection.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born in SMRU antenatal clinic, Maela camp
2. Written informed consent from the mother

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Maela is a densely populated camp predominantly inhabited by refugees of the Karen ethnic group. It is located in hills adjoining the Burmese border 50 km north of Mae Sot. It is the largest of the camps on the Thai-Burmese border, housing around one-third of the total refugee population. Maela has a population of approximately 43,000 people, of which 20% are females of child bearing age. Women presenting for antenatal care at SMRU's clinic will be asked to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD, Principal Investigator — Shoklo Malaria Research Unit
Locations (2):
- Thailand (2):
  - Shoklo Malaria Research Unit, MaeSod, Changwat Tak
  - Shoklo Malaria Research Unit, MaeSod